CLINICAL TRIAL: NCT06503991
Title: Community and Physician Perceptions of Barriers to Care for Acute Coronary Syndrome Among HIV-infected and -Uninfected Patients in Moshi, Tanzania_1
Brief Title: Acute Coronary Syndrome KCMC_1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00090902_1
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; HIV
MeSH Terms: conditions — Hypertension | interventions — Community Health Workers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COBRA and CHAMP (COACH) adapted intervention (Experimental): Persons living with HIV (PLWH) and receiving routine HIV care in northern Tanzania will receive an integrated COBRA (Control of Blood Pressure and Risk Attenuation) and CHAMP (Community Health Worker-delivered Hypertension Management Pilot) multi-component hypertension intervention.
  Interventions: Behavioral: Community Health Worker (CHW)-delivered Hypertension Management Pilot (CHAMP); Behavioral: Control of Blood Pressure and Risk Attenuation (COBRA)

INTERVENTIONS:
Behavioral: Community Health Worker (CHW)-delivered Hypertension Management Pilot (CHAMP) — Clinic-based hypertension educational intervention delivered by a Community Health Worker.
Behavioral: Control of Blood Pressure and Risk Attenuation (COBRA) — Multi-component counseling program addressing patient education, provider training, coordination of care, and subsidizing care costs.

SUMMARY:
To adapt and assess the implementation and preliminary effectiveness of an integrated COBRA and CHAMP multi-component community health worker-delivered hypertension intervention in improving blood pressure control among PLWH in northern Tanzania.

DETAILED DESCRIPTION:
Adapt and assess feasibility and preliminary effectiveness of an adapted community health worker-delivered hypertension intervention (Specific Objective 6): Using the ADAPT-ITT model, an interdisciplinary team of stakeholders will help adapt the COBRA intervention for integration within the HIV clinic to improve hypertension care among person living with HIV(PLWH) in Tanzania. The adapted, multicomponent, intervention (COACH) will integrate key components from our previous pilot intervention CHAMP with COBRA. The investigators anticipate the adapted intervention will include community health worker (CHW)-delivered hypertension counseling and blood pressure monitoring, integrated within existing HIV clinic appointments, referral to a prescribing provider within the HIV clinic for persistently elevated blood pressure, CHW-coordination and tracking of these referrals, provider training on use of an algorithmic protocol for blood pressure management, and subsidies to cover the unmet costs of antihypertensive agents. In the first 8 months, intervention content will be adapted using ADAPT-ITT. ADAPT-ITT is a pragmatic framework utilizing iterative, experiential processes to adapt evidence-based interventions. The investigators will assemble an inter-disciplinary Design Consultation Team (DCT) composed of key stakeholders who will participate in the intervention adaptation and design process which will occur iteratively through twice-monthly meetings between the study team and DCT. The DCT will include purposively selected patients with HIV and hypertension, clinicians and scientists from the US and Tanzania, clinic administrators, and community health workers. The investigators will document adaptation using the ADAPT-ITT framework.

Key staff, including community health workers, nurses, and physicians working at Majengo Care and Treatment Center (MCTC) and Pasua Care and Treatment Center (PCTC), will be trained with the final adapted COACH intervention, and this team will be responsible for implementing COACH in MCTC and PCTC. The investigators will then conduct a single arm pre-post feasibility study of COACH with 100 hypertensive participants recruited from MCTC and PCTC to determine implementation (reach, adoptability, implementation, and maintenance) and preliminary effectiveness outcomes (blood pressure, antihypertensive adherence, body mass index, waist circumference, CVD risk score, and hypertension knowledge) of the adapted intervention. Community health workers will measure blood pressure at initial enrollment and at monthly follow-up at HIV clinic and also participants with persistently elevated blood pressure at monthly follow-up. Any participant with SBP>=160mmHg and DBP>=100mmHg at enrollment will be referred to the hypertension coordinator and physician to be prescribed anti-hypertensives according to the COACH treatment algorithm. Participants with persistently elevated blood pressure (SBP ³140mmHg or DBP ³90mmHg) at 3- or 6- month follow-up will also be referred for pharmacotherapy. The investigators will compare participant blood pressure, antihypertensive adherence, body mass index, waist circumference, NHANES CVD risk score20 and hypertension knowledge (via the Hypertension Knowledge Level Scale21) at baseline and after six months of the intervention. The investigators will use quantitative and qualitative methods guided by the RE-AIM framework22to understand contexts of implementation of the adapted intervention. The investigators will use simple descriptive statistics to assess measures of reach and feasibility (i.e. the percentage of eligible MCTC and PCTC patients who enroll and the percentage of enrolled participants who 1) attend scheduled CHW visits; 2) are referred to a prescribing provider; 3) attend a referral appointment; 4) are prescribed anti-hypertensives; 5) report adherence to anti-hypertensives at 6-month follow up, and 6) the proportion of prescribed anti-hypertensives that conform to the COACH treatment algorithm. To assess adoption and acceptability of the intervention the investigators will conduct approximately 18 exit in-depth interviews with a subset of participants enrolled in COACH and also conduct approximately one - two focus group discussion with physicians, nurses, CHWS, and administrators to determine barriers and facilitators of intervention adoption and also resources, strategies and policies needed for intervention sustainability. To assess fidelity (i.e. the proportion of intervention components successfully delivered as designed) the investigators will audio record and review approximately 20% of CHW-delivered counseling to assess session completion and CHWs will complete a COACH fidelity checklist for each session.

ELIGIBILITY:
Inclusion Criteria:

* Known HIV
* Hypertension with single reading of SBP=>160 mm Hg and /or DBP=>100mm Hg
* Two separate measurements of SBP => 140 mmHg and/or DBP=> 90 mmHg

Exclusion Criteria:

* No documented elevated blood pressure
* No HIV infection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Hertz, MD, Principal Investigator — Duke University
Locations (1):
- KCMC, Moshi, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Min Htike WY, Manavalan P, Wanda L, Haukila K, Mmbaga BT, Sakita FM, Zebedayo R, Gwasma F, Jafar T, Bosworth HB, Thielman NM, Hertz JT. Community Health Worker Optimization of Antihypertensive Care in HIV (COACH): Study protocol for a pilot trial of an intervention to improve hypertension care among Tanzanians with HIV. PLoS One. 2024 Dec 17;19(12):e0315027. doi: 10.1371/journal.pone.0315027. eCollection 2024. PMID 39689146

RESULTS

PARTICIPANT FLOW:
Groups:
- COACH Intervention: Persons living with HIV (PLWH) and receiving routine HIV care in northern Tanzania will receive an integrated multi-component hypertension intervention, Community Health Worker Optimization of Antihypertensive Care in HIV (COACH).
  COACH consists of clinic-based hypertension educational counseling delivered by a Community Health Worker, provider training, coordination of care, and subsidizing care costs.
Period: Overall Study
Arm/Group | COACH Intervention
Started | 100
Completed | 96
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- CHAMP Intervention: Persons living with HIV (PLWH) and receiving routine HIV care in northern Tanzania will receive an integrated multi-component hypertension intervention, Community Health Worker Optimization of Antihypertensive Care in HIV (COACH).
  COACH consists of clinic-based hypertension educational counseling delivered by a Community Health Worker, provider training, coordination of care, and subsidizing care costs.
Arm/Group | CHAMP Intervention
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 100
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 100
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Tanzania | 100

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Measured by the Number of Total Scheduled Intervention Sessions (CHW Counseling Sessions, Doctor's Visits, Phone Calls) Attended
Description: The primary measure of feasibility for this study will be the number of total scheduled intervention sessions (CHW counseling sessions, doctor's visits, phone calls) attended by the 100 study participants over the course of the 6-month intervention.
Time Frame: 6 months
Measure: Count of Units; unit: Scheduled sessions
Units Other Than Participants: Scheduled sessions
Arm/Group | COACH Intervention
Number analyzed (Participants) | 100
Number analyzed (Scheduled sessions) | 600
Scheduled sessions | 589

2. Secondary Outcome: Number of Participants Reporting Adherence to an Anti-hypertensive Medication at 6-month Follow-up
Time Frame: 6 months
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | COACH Intervention
Number analyzed (Participants) | 96
Participants | 91

3. Secondary Outcome: Number of Participants With Controlled Blood Pressure at 6-month Follow-up
Description: Controlled blood pressure (BP) is defined as systolic BP<140 mmHg and diastolic BP <90 mmHg.
Time Frame: 6 months
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | COACH Intervention
Number analyzed (Participants) | 96
Participants | 73

4. Secondary Outcome: Hypertension Knowledge-Level Scale (HK-LS) Scores at 6-month Follow-up
Description: The HK-LS is used to measure knowledge about hypertension among adults. It has 22 items with six sub-dimensions. The maximum score is 22 for the entire scale, 2 for "definition", 4 for "medical treatment", 4 for "drug compliance", 5 for "lifestyle", 2 for "diet", and 5 for "complications" sub-dimensions. A higher score indicates greater hypertension knowledge.
Time Frame: 6 months
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COACH Intervention
Number analyzed (Participants) | 96
score on a scale | 20.4 (2.0)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | COBRA and CHAMP (COACH) Adapted Intervention
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT06503991/Prot_SAP_001.pdf
  • Informed Consent Form (2024-11-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT06503991/ICF_000.pdf